CLINICAL TRIAL: NCT01268696
Title: Genetic Assessment of the Patients With Metabolic Syndrome in Polish Population
Brief Title: Genetic Assessment of the Patients With Metabolic Syndrome
Acronym: GENMetS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Department of Medical Biotechnology, Medical University of Lodz
Other Study IDs: RNN/202/10/KE
Record Dates: First submitted 2010-12-28; First posted 2010-12-31 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2010-12

CONDITIONS: Metabolic Syndrome
Keywords: diabetes; obesity; hypertension; dyslipidemia
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Obesity; Hypertension; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — the blood samples taken into EDTA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control group: healthy volunteers
- Metabolic group: Patients with metabolic syndrome

SUMMARY:
Metabolic syndrome is a combination of medical disorders that increase the risk of developing cardiovascular disease and diabetes. The exact mechanisms of the complex pathways of metabolic syndrome are not yet completely known. The pathophysiology is extremely complex and has been only partially elucidated. Most patients are older, obese, sedentary, and have a degree of insulin resistance. Stress can also be a contributing factor. The most important factors are:

weight, genetics, aging, sedentary lifestyle,excess caloric intake. In our study we will assess the role of some polymorphisms in the pathology of metabolic syndrome.

DETAILED DESCRIPTION:
Eligibility criteria to the study:

* patients with metabolic syndrome
* with written consent

ELIGIBILITY:
Inclusion Criteria:

* patients with metabolic syndrome according to IDF,AHA and NHLBI 2009

Exclusion Criteria:

* diabetes type 1
* cancer
* not consent
* steroid therapy
* alcohol or drug abuse
* chronic inflammatory disease
* pregnancy or lactation
* severe hypothyroidism
* immunosuppressive treatment
* operation or severe injury during the last month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with metabolic syndrome
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-08 (Estimated); Study Completion 2015-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tadeusz Pietrucha, prof., Study Chair — Department of medical biotechnology
Locations (1):
- Department of medical biotechnology Medical University of Lodz, Lodz, Poland